CLINICAL TRIAL: NCT06370819
Title: Investigation of the Effect of Impaired Renal Function on the Pharmacokinetics of Subcutaneously Administered NNC0519-0130 in Participants With Various Degrees of Renal Function
Brief Title: A Research Study Looking Into Blood Levels of the Medicine NNC0519-0130 in the Body in Participants With Normal or Reduced Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN9541-4923; U1111-1292-3441 (Other: Universal Trial Number); 2023-506381-32 (Other: EU CT Number)
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NNC0519-0130 (Experimental): Participants will receive single subcutaneous (s.c.) dose of NNC0519-0130.
  Interventions: Drug: NNC0519-0130

INTERVENTIONS:
Drug: NNC0519-0130 — NNC0519-0130 will be administered subcutaneously.

SUMMARY:
NNC0519-0130 is a new medicine to improve the treatment options for people living with type 2 diabetes and people with overweight. In this study one dose of NNC0519-0130 will be given and blood levels of NNC0519-0130 will be compared between people with reduced kidney function and people with normal kidney function. The study will last up to 52 days including a screening phase of up to 28 days prior to dosing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of non-childbearing potential, aged 18-75 years (both inclusive) at the time of signing the informed consent.
* Body mass index (BMI) between 20.0 and 39.9 kilogram per square metre (kg/m^2) (both inclusive) at screening.
* Meeting the pre-defined glomerular filtration rate (GFR) criteria using estimated GFR (eGFR) based on the chronic kidney disease epidemiology collaboration (CKD-EPI) Creatinine Equation (2021) adjusted for estimated individual body surface area (BSA) for any of the renal function groups:
* For participants with normal renal function: eGFR of greater than or equal to 90 millilitres per minute (mL/min)
* Stage 2: For participants with mild renal impairment: eGFR of 60-89 mL/min
* Stage 3: For participants with moderate renal impairment: eGFR of 30-59 mL/min
* Stage 4: For participants with severe renal impairment: eGFR of 15-29 mL/min not requiring dialysis
* Stage 5: For participants with kidney failure: eGFR of less than 15 mL/min and requiring dialysis treatment

Exclusion Criteria:

* Any disorder which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol.
* Presence or history of any clinically relevant respiratory, metabolic, renal, hepatic, cardiovascular, gastrointestinal, or endocrinological conditions (except conditions associated with renal impairment or kidney failure) as judged by the investigator.
* Use of drugs known to affect creatinine clearance including cephalosporin and aminoglycoside, antibiotics, flucytosine, cisplatin, cimetidine, trimethoprim, cibenzoline and nitrofurantoin within 14 days or 5 half-lives, whichever is greater, before planned dosing of the investigational medicinal product (IMP).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC)0-∞,NNC0519-0130,SD: Area under the NNC0519-0130 plasma concentration-time curve after a single dose in participants with normal function, and mild, moderate and severe impairment | From baseline (visit 2, day 1) until completion of the end-of-study visit (visit 9, day 22)
  Measured in hours* nanomoles per litre (h*nmol/L).

SECONDARY OUTCOMES:
Maximum concentration (Cmax),NNC0519-0130,SD: Maximum observed NNC0519-0130 plasma concentration after a single dose in participants with normal function, and mild, moderate and severe impairment | From baseline (visit 2, day 1) until completion of the end-of-study visit (visit 9, day 22)
  Measured in nanomoles per litre (nmol/L).
AUC0-∞,NNC0519-0130,SD: Area under the NNC0519-0130 plasma concentration-time curve after a single dose in participants with kidney failure | From baseline (visit 2, day 1) until completion of the end-of-study visit (visit 9, day 22)
  Measured in hours* nanomoles per litre (h*nmol/L).
Cmax,NNC0519-0130,SD: Maximum observed NNC0519-0130 plasma concentration after a single dose in participants with kidney failure | From baseline (visit 2, day 1) until completion of the end-of-study visit (visit 9, day 22)
  Measured in nanomoles per litre (nmol/L).
Number of adverse events | From time of dosing (visit 2, day 1) until end of study (visit 9, day 22)
  Number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com